CLINICAL TRIAL: NCT02129257
Title: Single-arm Phase II Study of Maintenance Therapy With Aflibercept After First-line Treatment With FOLFIRI Plus Aflibercept in Metastatic Colorectal Cancer Patients
Brief Title: Clinical Trial of Combination Chemotherapy With Aflibercept in Patients With Advanced Colorectal Cancer
Acronym: AMALTHEA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE 6A/13; 2013-002567-26 (EudraCT Number)
Record Dates: First submitted 2014-04-28; First posted 2014-05-02 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — aflibercept; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFIRI-AFLIBERCEPT (Experimental): Aflibercept 4 mg/kg administered over 1 hour on Day 1, followed by FOLFIRI regimen. Treatment will be repeated every 2 weeks. FOLFIRI regimen: Irinotecan 180 mg/m² intravenous (IV) infusion and folinic acid 400 mg/m² IV infusion followed by: 5-fluorouracil (5-FU) 400 mg/m² IV bolus followed by: 5-FU 2400 mg/m² continuous IV infusion over 46 hours. FOLFIRI administration will immediately follow the aflibercept one. In the absence of PD after 6 months of the combination of chemotherapy and aflibercept, the patient will be treated with a maintenance therapy with aflibercept alone until PD or unacceptable toxicities, investigator's decision or patient's refusal of further treatment or death, whichever comes first.
  Interventions: Drug: AFLIBERCEPT; Drug: Irinotecan; Drug: 5-Fluorouracil; Drug: Folinic Acid

INTERVENTIONS:
Drug: AFLIBERCEPT
  Other Names: Zaltrap; AVE005
Drug: Irinotecan
  Other Names: Campto
Drug: 5-Fluorouracil
Drug: Folinic Acid

SUMMARY:
The AMALTHEA (Aflibercept MAintenance after first-Line THErapy with FOLFIRI+Aflibercept in metastatic colorectal cancer patients) trial is an investigator-initiated, single arm, open-label, phase II study. Patients with histologically proven metastatic colorectal carcinoma will be treated with a combination of FOLFIRI and aflibercept for 6 months. Both Kirsten rat sarcoma viral oncogene homolog (KRAS) wild type (wt) and mutant (mut) patients wil be enrolled. In the absence of Progressive Disease (PD) after 6 months of the combination of chemotherapy and aflibercept, the patient will be treated with a maintenance therapy with aflibercept alone until PD or unacceptable toxicity, investigator's decision or patient's refusal of further treatment or death, whichever comes first.

DETAILED DESCRIPTION:
Statistical hypotheses and sample size calculation:

It is estimated that the progression-free survival (PFS) rate at 1year will be improved from 33% (corresponding to a median PFS of 7.5 months [null hypothesis]) to 47% (corresponding to a median PFS of 11 months [alternative hypothesis]) with the combination of first-line Folinic acid/5-Fluorouracil/Irinotecan (FOLFIRI) plus aflibercept therapy in patients with metastatic colorectal cancer (mCRC). Using the one-stage Fleming's design, in order to reject the null hypothesis in a one-sided test with a type I error of 5% and power 80%, 73 patients will be needed to enter the study.

Analysis population:

* Intent-to-treat (ITT) population: all patients who will have given their informed consent and who will have been correctly registered to the study
* Evaluable population for tumor response: all treated patients, without major protocol deviation, with at least one tumor evaluation while on treatment (except for early disease progression or death) and evaluable for response
* Safety population: the subset of the ITT population that took at least one dose of study medication

Primary analysis:

The primary efficacy parameter will be PFS rate at 1 year and it will be calculated in the ITT population.

Analysis of secondary endpoints:

Response to treatment will be described in a frequency table along with the corresponding percentages and 95% exact confidence intervals.

Kaplan-Meier method will be used to estimate median PFS and overall survival (OS) values and 95% confidence intervals. All of these analyses will be performed in the ITT population. Analysis for objective response rate (ORR) will additionally be presented in the evaluable population for tumor response.

Adverse Events (AEs) of the safety population for the FOLFIRI-aflibercept treatment part and the maintenance therapy will be presented in frequency tables according to grade, along with the corresponding percentages (N, %).

Exploratory endpoints:

Univariate and multivariate Cox regression analyses will also be performed to explore prognostic factors among basic clinicopathological characteristics and evaluated biomarkers, with respect to PFS and OS. Time-to-event distributions for the expression of examined markers will be estimated by Kaplan-Meier method and compared using log-rank test.

Formalin-fixed embedded tumor tissue blocks will be collected from the primaries or metastases for the immunohistochemical and messenger ribonucleic acid (mRNA) study of key angiogenic effectors and regulators, such as: vascular endothelial growth factor A (VEGF A), vascular endothelial growth factor A-121 (VEGFA-121), vascular endothelial growth factor A121b (VEGFA121b), short and long VEGFA isoforms, metalloproteinase inhibitor 3 (TIMP3), vascular endothelial growth factor B (VEGF-B), placental growth factor (PlGF), vascular endothelial growth factor-C (AVEGF-C), Semaphorins, hypoxia-inducible factor 1 (HIF1), vascular endothelial growth factor receptor 1 (VEGFR1), vascular endothelial growth factor receptor 2 (VEGFR2), neuropilin 1 (NRP1), neuropilin 2 (NRP2), thrombospondin 1 (TSP1), thrombospondin 2 (TSP2), angiopoietin-1 (Ang1), Angiopoietin-2 (Ang2), Tie2, interleukin 8 (IL8), CXC chemokine receptor 1 (CXCR1), CXC chemokine receptor 2 (CXCR2)

Pharmacokinetic(PK)/Pharmacodynamic analyses (PD) PK/PD assessments (plasma analytes, plasma free and VEGF-bound aflibercept) will be performed in all registered and treated patients at specified timepoints during both FOLFIRI-aflibercept induction and aflibercept maintenance therapy, to assess the free/bound aflibercept ratio over cycles and the potential correlation with clinical endpoints (safety and efficacy).

ELIGIBILITY:
Inclusion Criteria

* Histologically proven adenocarcinoma of the colon and/or rectum
* Metastatic disease confirmed clinically/radiologically
* Signed written informed consent
* No prior therapy for metastatic disease
* Duly documented inoperable metastatic disease, ie not suitable for complete curative surgical resection
* At least one measurable or evaluable lesion as assessed by Computed Tomography (CT) scan or MRI (Magnetic Resonance Imaging) according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) Performance status (PS) 0-2
* Adequate hematological status:

  * neutrophils (ANC) ≥1.5x109/L
  * platelets ≥100x109/L
  * haemoglobin ≥9g/dL
* Adequate renal function: serum creatinine level <1.5 mg/dl and Glomerular Filtration Rate>50 ml/min by Cockroft/Gault formula
* Adequate liver function:

  * serum bilirubin ≤1.5 x upper normal limit (ULN)
  * alkaline phosphatase
  * aspartate aminotransferase (AST)
  * alanine aminotransferase (ALT) < 5 x ULN
* Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour
* Regular follow-up feasible
* Baseline evaluations performed before registration: clinical and blood evaluations no more than 2 weeks (14 days) prior to registration, tumor assessment (chest X-ray, CT-scan or MRI, evaluation of non-measurable lesions) no more than 3 weeks (21 days) prior to registration
* First course of treatment planned less than 1 week (7 days) after registration
* For female patients of childbearing potential, negative serum pregnancy test within 1 week (7 days) prior of starting study treatment
* Female patients must commit to using reliable and appropriate methods of contraception until at least three months after the end of study treatment (when applicable). Male patients with a partner of childbearing potential must agree to use contraception in addition to having their partner use another contraceptive method during the trial.

Exclusion Criteria

* Exclusive presence of bone metastasis only
* Uncontrolled hypercalcemia
* Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg despite medical therapy), or history of hypertensive crisis, or hypertensive encephalopathy
* Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy)
* Treatment with any other investigational medicinal product within 28 days prior to study entry
* Other serious and uncontrolled non-malignant chronic disease
* History or presence of Central Nervous System (CNS) metastasis unless adequately treated (e.g. non irradiated CNS metastasis, seizures not controlled with standard medical therapy)
* Gilbert's syndrome
* Intolerance to atropine sulfate or loperamide
* Known dihydropyrimidine dehydrogenase deficiency
* Treatment with Cytochrome P450 3A4 (CYP3A4) inducers unless discontinued > 7 days prior to randomization
* Any of the following in 3 months prior to inclusion: grade 3-4 gastrointestinal bleeding (unless due to resected tumor), treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, or diverticulitis
* Other concomitant or previous malignancy, except:

  * adequately treated in-situ carcinoma of the uterine cervix
  * basal or squamous cell carcinoma of the skin
  * cancer in complete remission for >5 years
* Any other serious and uncontrolled non-malignant disease, major surgery or traumatic injury within the last 28 days
* Pregnant or breastfeeding women
* Patients with known allergy to any excipients to study drugs
* History of myocardial infarction and/or stroke or other arterial thrombotic events or pulmonary embolism or unstable angina pectoris within 6 months prior to registration
* Poorly controlled cardiac arrhythmias
* Bowel obstruction
* History of severe tumour bleeding or bleeding disorders
* Poorly controlled anti-coagulation therapy (INR>3.0 on coumadin or heparin compounds)
* Palliative radiation therapy within 4 weeks prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-05-26 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) rate at 1 year | Up to 1 year

SECONDARY OUTCOMES:
Evaluation of Objective Response Rate (ORR) defined as the proportion of patients with complete response (CR) or partial response (PR) among all patients, as assessed according to Response Evaluation Criteria for Solid Tumors (RECIST) v1.1 | Up to 20 months
  Response to treatment will be described in a frequency table along with the corresponding percentages and 95% exact confidence intervals.
Evaluation of Overall Survival (OS) | Time interval from registration to the date of death due to any cause assessed up to 60 months
Evaluation of Progression-Free Survival (PFS) | Time interval from registration to the first date of documented progression or death due to any cause assessed up to 60 months
Number of participants with Serious and Non-Serious Adverse Events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 | Up to 40 months
  Adverse Events of the safety population for the FOLFIRI-aflibercept treatment part and the maintenance therapy will be presented in frequency tables according to grade, along with the corresponding percentages (N,%)
Tumor tissue mRNA levels of VEGFA-121, VEGFA121b, VEGF-B, PlGF, VEGF-C, Semaphorins, HIF1, VEGFR1, VEGFR2, Neuropilins 1,2, Thrombospondin, Angiopoietins 1,2. Predictive significance for response rate, PFS, OS. | Tumor blocks will be collected at baseline
Steady-state concentration of free Aflibercept and VEGF-bound Aflibercept in plasma. Predictive significance for response rate, PFS, OS. | On day 1 of cycle 1, on day 1 of cycle 3, on day 1 of week 3 of Aflibercept maintenance monotherapy, at the end of treatment, assessed up to 20 months
Enzyme-linked immunosorbent assay (ELISA) plasma concentrations of VEGFA, soluble VEGFR1, soluble VEGFR2, VEGF-B, PlGF, basic fibroblast growth factor (bFGF), hepatocyte growth factor (HGF). Predictive significance for response rate, PFS, OS. | On day 1 of cycle 1, on day 1 of cycle 3, on day 1 of week 3 of Aflibercept maintenance monotherapy, at the end of treatment, assessed up to 20 months

CONTACTS AND LOCATIONS:
Overall Officials: George Pentheroudakis, MD, Ass.Prof, Study Chair — Dept of Medical Oncology, Ioannina University Hospital
Locations (18):
- Greece (18):
  - Agios Georgios Chania General Hospital, Chania, Mournies
  - 2nd Dept of Internal Medicine, Agios Savvas Cancer Hospital, Athens
  - 251 Airforce Hospital, Athens
  - 2nd Dept of Internal Medicine, General Hospital of Athens "Hippokratio", Athens
  - Oncology Unit, 3rd Dept of Internal Medicine, Athens School of Medicine, Sotiria General Hospital, Athens
  - Oncology Section, Dept of Clinical Therapeutics, General Hospital of Athens "Alexandra", Athens
  - Division of Oncology, 2nd Dept of Internal Medicine, University Hospital "Attiko", Athens
  - 2nd Dept of Medical Oncology, Agii Anargiri Cancer Hospital, Athens
  - 3rd Dept of Medical Oncology, Agii Anargiri Cancer Hospital, Athens
  - 3rd Dept of Medical Oncology, Hygeia Hospital, Athens
  - 1st Dept of Medical Oncology, Metropolitan Hospital, Athens
  - 2nd Dept of Medical Oncology, Metropolitan Hospital, Athens
  - Dept of Medical Oncology, University Hospital of Heraklion, Heraklio
  - Dept of Medical Oncology, Ioannina University Hospital, Ioannina
  - Oncology Dept, University Hospital of Larissa, Larissa
  - Division of Oncology, Dept of Internal Medicine, University Hospital of Patras, Pátrai
  - Thermi Clinic S.A., Thermi
  - Dept of Medical Oncology, Papageorgiou General Hospital, Thessaloniki